CLINICAL TRIAL: NCT06238518
Title: Intravascular Lithotripsy Versus Conventional Therapy for Severely Calcified Coronary Artery Lesions: an Investigator-initiated, Open-label, Multicentre, Randomised, Superiority Trial
Brief Title: Intravascular Lithotripsy Versus Conventional Therapy for Severely Calcified Coronary Artery Lesions
Acronym: REC-CHIPCAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, LingTao, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20232390-C-1
Record Dates: First submitted 2024-01-16; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Severely Calcified Coronary Stenoses; De Novo Stenosis
Keywords: Severely Calcified Coronary Stenoses; Intravascular Lithotripsy; percutaneous coronary intervention

STUDY DESIGN:
Intervention Model Description: Prospective, 1:1 randomized, controlled, multicenter trial to assess effectiveness and safety of adding IVL to Conventional Therapy compared to Conventional Therapy only in calcified coronary lesions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional lesion preparation plus Intravascular Lithotripsy strategy (Experimental): IVL could be performed before, amidst, or after Conventional lesion preparation therapy; However, the use of IVL treatment is mandatory.
  Interventions: Procedure: Intravascular Lithotripsy; Procedure: Conventional lesion preparation strategy
- Conventional lesion preparation strategy (Active Comparator): Conventional lesion preparation strategy includes the use of Compliant, noncompliant, cutting, or scoring balloons, Excimer laser coronary atherectomy, or Rotational atherectomy at the discretion of the operator.
  Interventions: Procedure: Conventional lesion preparation strategy

INTERVENTIONS:
Procedure: Intravascular Lithotripsy — The size of the IVL balloon catheter is selected in a 1:1 ratio to the distal reference vessel diameter. The balloon catheter is then inflated to 4 atm, and 10 impulses are delivered. Subsequently, the balloon is inflated to 8 atm and then deflated to re-establish blood flow. Up to 100 impulses can be delivered, and the balloon can be repositioned within the lesion. In cases involving multiple lesions with different reference vessel diameters, various sizes of IVL balloons may be employed. If the IVL balloon catheter is unable to pass through the lesion, pre-dilatation can be performed using a smaller diameter noncompliant balloon or rotational atherectomy.
  Arms: Conventional lesion preparation plus Intravascular Lithotripsy strategy
Procedure: Conventional lesion preparation strategy — Conventional lesion preparation strategy includes the use of Compliant, noncompliant, cutting, or scoring balloons, Excimer laser coronary atherectomy, or Rotational atherectomy at the discretion of the operator.

SUMMARY:
Percutaneous coronary intervention (PCI) encounters challenges with calcified coronary lesions, leading to potential issues such as failed balloon dilatation, incomplete stent expansion, and increased risks of adverse events post-PCI, including stent restenosis and thrombosis.

Intravascular lithotripsy (IVL), a novel approach for severely calcified coronary lesion preparation, has shown promising preliminary outcomes. Combining IVL with conventional approaches, such as Rotational atherectomy (RA), non-compliant balloons, or cutting balloons, may associated with additional benefit than conventional approaches only in terms of better stent expansion and lower long-term adverse events.

This pilot randomized trial aims to investigate whether combining IVL to conventional therapy surpasses the efficacy of conventional approaches alone. The primary effectiveness endpoint is final stent expansion assessed by post-procedure optical coherence tomography (OCT), and the primary safety endpoint is target lesion failure (TVF). The trial seeks to provide valuable insights into the optimal approach for managing severely calcified coronary lesions during PCI.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. Patients with acute or chronic coronary artery syndrome indicated for PCI with stenting.
2. Able to understand and provide informed consent and comply with all study procedures

Angiographic Inclusion Criteria:

1. Native and de novo coronary artery disease
2. Lesion navigable by a 0.014" guidewire.
3. Target lesion is severely calcified, meeting one of the following criteria:

   * Presence of calcium ≥ 270°, lengths ≥ 5mm, and thickness ≥ 0.5mm at one cross-section as assessed by OCT
   * If the OCT catheter is unable to pass through the target lesion after dilatation due to calcification or tortuosity, and the target lesion is severely calcified on both sides of the arterial wall during angiography, with the length of the calcification >15 mm, the lesion will be recognized as a severely calcified lesion, meeting the criteria for enrollment

Exclusion Criteria:

General Exclusion Criteria:

1. Patients under 18 years of age.
2. Incapable of providing informed consent.
3. Female patients who are pregnant or nursing (a pregnancy test must be conducted within 7 days before the index procedure for women of childbearing potential, as per local practice).
4. Concurrent medical conditions with a life expectancy of less than 1 year.
5. Hemodynamic instability.
6. Known contraindications to medications such as Heparin, anticoagulation, antiplatelet drugs, or contrast.
7. Active bleeding.
8. New-onset stroke or transient ischemic attack (TIA) within 90 days prior to enrollment.
9. Severe renal dysfunction (eGFR ≤ 30 ml/min).
10. Patients scheduled to undergo cardiac intervention or cardiac surgery within 30 days of the index procedure.
11. Recent ST-segment elevation myocardial infarction (STEMI) within 7 days or recent cardiogenic shock.
12. Lesions located in surgical conduits.

Angiographic Exclusion Criteria:

1. Target vessel exhibiting C-F type dissection.
2. Thrombosis observed by angiography or OCT.
3. Presence of an aneurysm within 10 mm of the target lesion.
4. Left main ostial lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Final stent expansion (%) assessed by OCT | Measured by the data collected at the end of the PCI procedure
  The primary efficacy endpoint of the trial is the Final stent expansion %, defined as the minimum stent area (MSA) / mean reference lumen area assessed by OCT.
Target vessel failure (TVF) | 1, 12, 36, and 60 months
  The primary safety endpoint of the trial is target vessel failure (TVF), defined as a non-hierarchical composite endpoint of cardiovascular death, target-vessel myocardial infarction (TV-MI), and clinically indicated target vessel revascularization (CI-TVR).

SECONDARY OUTCOMES:
Major cardiovascular adverse events | 1, 12, 36, and 60 months
  Major adverse cardiovascular events (MACE) is defined as a hierarchical composite of cardiovascular death, target-vessel myocardial infarction, clinically indicated target vessel revascularization, stent delivery failure, and suboptimal stent deployment.
  The between-group difference in terms of MACE will be compared using the Win Ratio approach in the abovementioned order.

OTHER OUTCOMES:
Suboptimal stent deployment | Measured by the data collected at the end of the PCI procedure
  Suboptimal stent deployment is defined as fulfilling any of the following criteria: minimum stent area (MSA) ≤4.5mm2 (by OCT), MSA/mean reference lumen area ≤80%, flow-limiting dissections, or incomplete stent apposition (axial distance ≥0.4 mm and length ≥1 mm)
Stent delivery failure | Measured by the data collected at the end of the PCI procedure
Cardiac cause death | 1, 12, 36, and 60 months
Target vessel myocardial infarction (TV-MI) | 1, 12, 36, and 60 months
Clinically indicated target lesion revascularization (CI-TLR) | 1, 12, 36, and 60 months
Clinically indicated target vessel revascularization (CI-TVR) | 1, 12, 36, and 60 months
All cause death | 1, 12, 36, and 60 months
Any stroke | 1, 12, 36, and 60 months
Any MI | 1, 12, 36, and 60 months
Any revascularisation | 1, 12, 36, and 60 months
Patient-oriented composite endpoint (PoCE) | 1, 12, 36, and 60 months
  Patient-oriented composite endpoint (PoCE) is defined as all-cause death, any stroke, any MI, and any clinically indicated revascularisation
Definite/Probable Stent thrombosis rates | 1, 12, 36, and 60 months
  According to ARC-II classification
Peri-procedural MI | 48 hours
  According to SCAI definition
Peri-procedural major adverse events | 30 days
  Peri-procedural major adverse events were defined as a composite of the procedure of periprocedural MI, flow-limiting dissections, perforation/rupture, acute occlusion, slow-flow/no-reflow, ventricular tachycardia/ventricular fibrillation within 30 days
Acute gain | Measured by the data collected at the end of the PCI procedure
  Acute gain is the difference between post- and pre-procedural minimal lumen diameter (MLD) as measured in (preferable) identical orthogonal views by OCT (MLDpost - MLDpre)
The difference between post- and pre-procedural FFR/IMR | Measured by the data collected at the end of the PCI procedure
  FFR/IMR can be measured either by wire or derived from coronary angiography
Procedure time of the PCI | Measured by the data collected at the end of the PCI procedure
Radiation dose of the PCI | Measured by the data collected at the end of the PCI procedure
Contrast volume | Measured by the data collected at the end of the PCI procedure
Calcium fracture | Measured by the data collected at the end of the PCI procedure
Angiographic success | Measured by the data collected at the end of the PCI procedure
  Angiographic success is defined as the ability of the allocated treatment to produce residual stenosis <20% after stenting without serious angiographic complications (severe dissection impairing flow [type D-F], perforation, abrupt closure, persistent slow flow, or no-reflow).
Strategy success | Measured by the data collected at the end of the PCI procedure
  Strategy success is defined as Angiographic success without treatment crossover or stent loss
Clinical (Procedural) success | 1 month
  Clinical (Procedural) success is defined as Device success without the occurrence of in-hospital cardiovascular death, target-vessel myocardial infarction, or clinically indicated target vessel revascularization.
Coronary flow velocity | Measured by the data collected at the end of the PCI procedure
  Coronary flow velocity is measured by Quantitative Flow Ratio (QFR)
TIMI Flow | Measured by the data collected at the end of the PCI procedure
Stent malapposition | Measured by the data collected at the end of the PCI procedure
Stent volume / reference lumen volume | Measured by the data collected at the end of the PCI procedure
  Assessed by OCT
Mean stent area / Mean reference lumen area | Measured by the data collected at the end of the PCI procedure
  Assessed by OCT Assessed by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D, Ph.D., Study Chair — Xijing Hospital; Chao Gao, M.D, Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China